CLINICAL TRIAL: NCT00227344
Title: Catheter Ablation for Cure of Atrial Fibrillation
Brief Title: CACAF2 Study: Catheter Ablation for Cure of Atrial Fibrillation
Acronym: CACAF-2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study prematurely terminated due to randomization imbalance.
Sponsor: Biosense Webster EMEA (Industry)
Responsible Party: Sponsor
Organization: Biosense Webster, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACAF2
Record Dates: First submitted 2005-09-15; First posted 2005-09-28 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Catheter ablation
  Interventions: Device: RF ablation
- 2 (Active Comparator): Antiarrhythmic drugs
  Interventions: Drug: Antiarrhythmic drugs

INTERVENTIONS:
Device: RF ablation — Catheter ablation with NAVISTAR® THERMOCOOL® Catheter in conjunction with CARTO™ EP Navigation System
  Arms: 1
Drug: Antiarrhythmic drugs — Best antiarrhythmic drug according to local practice (amiodarone suggested) throughout the study
  Arms: 2

SUMMARY:
The objective of this prospective multicenter randomized study is to establish the effectiveness of treatment of persistent atrial fibrillation by encircling the pulmonary veins with radiofrequency (RF) ablation and creating additional lines of block with the aid of the NAVISTAR® THERMOCOOL® catheter in conjunction with the CARTO™ EP Navigation System. Effectiveness will be determined by comparing the chronic success of ablation therapy versus antiarrhythmic drug therapy, defined as the absence of persistent tachyarrhythmias during the first 24 months after a run-in phase of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* Written informed consent
* One documented relapse of atrial fibrillation (AF) during antiarrhythmic drug therapy after an electrical cardioversion

Exclusion Criteria:

* Permanent atrial fibrillation
* Patients who had tried >1 antiarrhythmic drug (Class I or Class III).
* AF was the sole rhythm for >6 months before the enrollment.
* Previous ablation for AF.
* AF is deemed secondary to a transient or correctable abnormality including electrolyte imbalance, trauma, recent surgery, infection, toxic ingestion, and endocrinopathy.
* Patients who have fibrillation episodes triggered by another uniform arrhythmia (eg, atrial flutter or atrial tachycardia).
* Patients with intra-atrial thrombus, tumor, or another abnormality that precludes catheter introduction.
* Patients with Wolf-Parkinson-White syndrome.
* Patients awaiting cardiac transplantation.
* Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-III-IV or ejection fraction (EF) <40%.
* Patients with unstable angina or acute myocardial infarction within 3 months.
* Patients with cardiac revascularization or other cardiac surgery within 6 months.
* Patients with heart disease in which corrective surgery is anticipated.
* Patients in whom appropriate vascular access is precluded.
* Pregnant women.
* A separate requirement for antiarrhythmic drug treatment, which will require an antiarrhythmic drug not previously tried for AF suppression.
* Prior atrial surgery.
* Contraindication to treatment with warfarin or other bleeding diathesis.
* Renal failure requiring dialysis.
* Hepatic failure.
* Participant in investigational clinical or device trial.
* Unwilling or unable to give informed consent.
* Inaccessible for follow-up.
* Psychological problem that might limit compliance.
* Active abuse of alcohol or other drugs which may be causative of AF.
* An implanted device (pacemaker or cardioverter-defibrillator).
* Left atrial diameter (anteroposterior) >50 mm.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2004-12; Primary Completion 2008-10 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Bertaglia, MD, Principal Investigator — ULSS n.13, Mirano (VE), Italy; Giuseppe Stabile, MD, Principal Investigator — Casa di Cura San Michele, Maddaloni, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred twenty-nine (129) subjects were enrolled in the study at the time of termination. Ten of 13 study sites were in Italy, thus the majority of subjects were recruited from Italian sites. The sponsor's decision at study termination was to report primary and secondary endpoints for which meaningful data analysis was possible.
Groups:
- Catheter Ablation: Catheter Ablation
- Antiarrhythmic Drug Treatment: Best antiarrhythmic drug according to local practice (amiodarone suggested) throughout the study
Period: Overall Study
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Started | 87 | 42
Completed | 75 | 37
Not Completed | 12 | 5
Not completed — study terminated early | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment | Total
Number analyzed (Participants) | 87 | 42 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (8.9) | 64.3 (4.7) | 59.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 70 | 21 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Absence of Persistent Atrial Tachyarrhythmias Relapse During the First 24 Months After the run-in Phase (2 Months).
Description: Persistent atrial tachyarrhythmia is defined as lasting 7 or more days per two consecutive transtelephonic monitoring or electrocardiogram recordings (obtained at least one week apart) with no cardioversions.
Time Frame: within first 24 months after a 2-month run-in phase
Population: Intention to treat (ITT) analysis includes subjects with available transtelephonic monitoring data.
Measure: Number; unit: percentage of participants
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Number analyzed (Participants) | 75 | 37
percentage of participants | 36.0 | 45.9

2. Secondary Outcome: Percentage of Participants With Total Absence of Any Documented Atrial Tachyarrhythmias Lasting Longer Than 30 Seconds During the First 24 Months After the run-in Phase (2 Months)
Time Frame: within first 24 months after a 2-month run-in phase
Population: Intention to treat (ITT) analysis includes subjects with available transtelephonic monitoring data.
Measure: Number; unit: percentage of participants
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Number analyzed (Participants) | 75 | 37
percentage of participants | 16.0 | 24.3

3. Secondary Outcome: Percentage of Procedural Success
Description: Procedural success was determined on the day of the procedure (Day 0) and was based on responses to the following:
  1. "Has a validation of the lesions been performed by taking 3 points inside each circular lesion?"
  2. "If YES to #1, did you observe that none of them exceed 0.1 mV?"
  3. "Did you observe any adverse event during the procedure?"
  If the answers to (1 ) and (2 ) were YES and (3) was NO, then the procedure was determined a success.
Time Frame: The day of the procedure
Population: Procedural success was only calculated for the catheter ablation group. Intention to Treat (ITT) analysis of procedural success for the catheter ablation group was performed using available data. The "0" below the Antiarrhythmic Drug treatment group represents "not available."
Measure: Number; unit: percentage of participants
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Number analyzed (Participants) | 84 | 0
percentage of participants | 70.2 |

4. Secondary Outcome: Time to First Recurrence of Any Tachyarrhythmias Lasting 30 or More Seconds After the Run in Phase
Time Frame: day 61 through 790
Population: Intention to treat (ITT) analysis includes subjects with available transtelephonic monitoring data. The upper bound of the confidence interval for the drug treatment group could not be calculated because of the high censoring rate. Therefore, "NA" is more appropriate in place of the maximum duration of follow-up (790.0) as the upper bound.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Number analyzed (Participants) | 75 | 36
days | 302.0 [133.0 to 436.0] | 328.0 [165.0 to NA] — The upper bound of the confidence interval for the drug treatment group could not be calculated because of the high censoring rate. Therefore, "NA" is more appropriate in place of the maximum duration of follow-up (790.0) as the upper bound.

5. Secondary Outcome: Percentage of Participants Achieving Clinical Success (Subjects Taking AADs That Remain Free From Any Tachyarrhythmias) in Association With Antiarrhythmic Drugs
Time Frame: at 26 months and at each patients last follow-up visit
Population: Study termination due to randomization imbalance. Data not analyzed since enrollment limited and therefore insufficient data to identify meaningful differences and draw significant conclusions. The "0" below represents "not available."
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quality of Life
Time Frame: at 14, 26 and 38 months
Population: as for outcome 5
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Health-economics Parameters (Days of Hospitalization)
Time Frame: at 26 months and at each patients last follow-up visit
Population: Data not analyzed due to study termination - insufficient data to identify meaningful differences and draw significant conclusions.
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants With Normal Sinus Rhythm at the Last Follow-up Visit Measured by ECG and 24-hour Holter Monitor
Time Frame: at each patients last follow-up visit
Population: Intention to Treat (ITT)analysis of sinus rhythm was performed for subjects with available Holter Monitor data.
Measure: Number; unit: percentage of participants
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Number analyzed (Participants) | 82 | 39
percentage of participants | 75.6 | 51.3

ADVERSE EVENTS:
Arm/Group | Catheter Ablation | Antiarrhythmic Drug Treatment
Serious Adverse Events (participants affected / at risk) | 25/87 | 22/42
Other Adverse Events (participants affected / at risk) | 0/87 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter Ablation (N=87) | Antiarrhythmic Drug Treatment (N=42)
coronary angiography (Cardiac disorders) | 0 (0) | 1 (1)
all types of atrial flutter including, but not limited to atypical and left atrial flutter (Cardiac disorders) | 3 (3) | 1 (1)
worsening ventricular function (Cardiac disorders) | 0 (0) | 1 (1)
sinusal arrest (Cardiac disorders) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
heart failure (Cardiac disorders) | 2 (2) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
low hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
lipotimia and hyperkaliemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2)
reduced visual acuity secondary to cataract (Eye disorders) | 0 (0) | 1 (1)
sudden death (General disorders) | 0 (0) | 1 (1)
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
increased tumor size (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
tremens (Nervous system disorders) | 0 (0) | 1 (1)
renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ablate and pace procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
silent ischemic heart disease (Cardiac disorders) | 0 (0) | 1 (1)
carotid atrery stenosis (Vascular disorders) | 0 (0) | 1 (1)
sinus pause (Cardiac disorders) | 2 (2) | 0 (0)
dyspnea (Cardiac disorders) | 2 (2) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
diabetes (Endocrine disorders) | 1 (1) | 0 (0)
colon polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
cardiac tamponade (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
inguinal hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
cerebral aneurism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
right knee trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
brain injury secondary to facial trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
genital-urinary area neoplastic mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
nasal bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pacemaker implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
atrioventricular node ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
transient ischemic attack (Vascular disorders) | 1 (1) | 0 (0)
artero-venious fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter Ablation (N=87) | Antiarrhythmic Drug Treatment (N=42)
corneal deposit of amiodarone (Eye disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated early due to randomization imbalance. The relatively small number of subjects enrolled limited the amount of data available for analysis. Because the study did not reach its targeted enrollment, the study is underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.